CLINICAL TRIAL: NCT05439330
Title: Application of a Dental-dedicated MRI in the Diagnosis of Temporomandibular Joint Disorders, Tissue Alterations Related to Third Molars, Periapical and Periodontal Inflammatory Diseases, and Implant Planning
Brief Title: Application of a Dental-dedicated MRI in the Diagnosis of Temporomandibular Joint Disorders, Tissue Alterations Related to Third Molars, Periapical and Periodontal Inflammatory Diseases, and Implant Treatment Planning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry); Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Jennifer Christensen, DDS, ph.d., University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91340
Record Dates: First submitted 2022-06-20; First posted 2022-06-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: TMJ; Apical Periodontitis; Periodontal Inflammation; Retained Tooth; MRI
MeSH Terms: conditions — Periapical Periodontitis; Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: Each person has a MRI scan done following the requested radiograph. MRI and radiographs are compared for diagnostic purposes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of a dental-dedicated MRI (Experimental): MRI of conditions related to teeth and surrounding structures
  Interventions: Device: MRI of teeth and surrounding structures

INTERVENTIONS:
Device: MRI of teeth and surrounding structures — included above

SUMMARY:
The aim of the present study is to show that the use of 0.55T MRI combined with a "dental" coil produces images of sufficient diagnostic value to assess areas of interest in dentistry, and to compare MR images to traditional, dental-oriented radiographic images for diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria (one of the following):

* referred for CBCT imaging of at least one tooth for endodontic reasons
* referred for intra-oral and/or panoramic imaging covering at least one molar tooth for periodontal reasons
* referred for CBCT imaging of the TMJ (bilaterally)
* referred for panoramic imaging of the third molar (retained/semi-retained, uni- or bilateral), prior to treatment planning
* referred for CBCT imaging prior to implant treatment

Exclusion Criteria:

* younger than 18 years
* unable to give consent
* pregnant
* pronounced claustrophobia
* pacemakers or implanted defibrillators
* metal shrapnel injuries of the eyes or MRI incompatible metallic inclusions or implants large tatoos
* non-removable piercings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Application of a dental-dedicated MRI in the diagnosis of temporomandibular joint disorders, tissue alterations related to third molars, periapical and periodontal inflammatory diseases, and implant treatment planning | 2½ years
  Diagnosis of pathologies in the TMJ (e.g. disc displacement (anterior/posterior/lateral), inflammation (yes/no), bone changes (yes/no)), periodontal defects (e.g. bone defects (mm), inflammation (yes/no)), periapical pathology (e.g. inflammation (yes/no), apical periodontitis (yes/no)), bone measurements in edentulous areas, and third molars (e.g. relation to surrounding structures (over/same level/under nerve), resorption of neighboring teeth (yes/no)) seen on MRI compared to diagnosis obtained in radiographs. Observations seen on MRI will be compared to observations seen in radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Spin-Neto, ph.D, Study Chair — University of Aarhus
Locations (1):
- IOOS, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No